CLINICAL TRIAL: NCT03206060
Title: Lu-177-DOTATATE (Lutathera) in Therapy of Inoperable Pheochromocytoma/ Paraganglioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170087; 17-C-0087
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: Pheochromocytoma; Paraganglioma; Neuroendocrine Tumors; Neuroendocrine Neoplasms
Keywords: Hypertension; Catecholamine; Familial Syndromes; Somatostatin Receptors; Ionizing Radiation
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Neuroendocrine Tumors; Hypertension | interventions — lutetium Lu 177 dotatate; gallium Ga 68 dotatate; amino-acid, glucose, and electrolyte solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Lu-177-DOTATATE (Experimental): Lu-177-DOTATATE is administered IV every 8 (+/- 2) weeks, for a total of 4 administrations. A Ga-68-DOTATATE PET and F-18-FDG-PET, as well as CT/ MRI for RECIST monitoring, will be obtained post 2 administrations and post 4 administrations. Concomitant administration of an IV infusion of an amino acid (AA) solution will also be done for renal protection. Concomitant administration of an IV infusion of an amino acid (AA) solution will also be done for renal protection.
  Interventions: Drug: Lu-177-DOTATATE; Drug: Ga-68-DOTATATE; Drug: F-18-FDG; Drug: Amino Acid solution

INTERVENTIONS:
Drug: Lu-177-DOTATATE — Lu-177-DOTATATE IV at weeks 1, 8, 16 and 24.
Drug: Ga-68-DOTATATE — Ga-68-DOTATATE PET/CT at weeks 15 and 31, every 24 weeks during 3 years follow up period.
Drug: F-18-FDG — F-18-FDG PET/CT at weeks 15 and 31, every 24 weeks during 3 years follow up period.
Drug: Amino Acid solution — AA solution will be administered 60 minutes prior to each Lu-177-DOTATATE infusion.

SUMMARY:
Background:

Pheochromocytoma and paraganglioma are rare tumors. They usually form inside and near the adrenal gland or in the neck region. Not all these tumors can be removed with surgery, and there are no good treatments if the disease has spread. Researchers think a new drug may be able to help.

Objective:

To learn the safety and tolerability of Lu-177-DOTATATE. Also, to see if it improves the length of time it takes for the cancer to return.

Eligibility:

Adults who have an inoperable tumor of the study cancer that can be detected with Ga-68-DOTATATE PET/CT imaging

Design:

Participants will be screened with a medical history, physical exam, and blood tests.

Eligible participants will be admitted to the NIH Clinical Center.

Participants will get the study drug in an intravenous infusion. They will get 4 doses, given about 8 weeks apart.

Between 4 and 24 hours after each study drug dose, participants will have scans taken. They will lie on their back on a scanner table.

Participants will have vital signs taken. They will give blood and urine samples.

During the study, participants will have other scans taken. Some scans will use a radioactive tracer.

Participants will complete quality of life questionnaires.

Participants will be contacted by phone 1-3 days after they leave the Clinical Center. They will then be followed every 3 to 6 months for 3 years or until their disease gets worse.

DETAILED DESCRIPTION:
Background:

* Pheochromocytomas/paragangliomas (PHEOs/PGLs) are rare tumors arising from neural crest tissue that can develop in sympathetic and parasympathetic paraganglia throughout the body. Those arising in the adrenal gland are called PHEOs while those located extra-adrenally are called PGLs.
* While benign and uni-focal, PHEO/PGL can be effectively treated with surgical resection, participants with metastatic PHEO/PGL often times have few effective and efficient treatment options with current treatments aimed more at palliation and symptom control. Furthermore, some benign head and neck PGLs may be inoperable because of their size and location.
* Somatostatin receptors (SSTR), especially type 2, have been shown to be over-expressed in a number of human tumors, including gastroenteropancreatic (GEP), carcinoids, neuroblastoma, prostate cancer, and PHEO/PGL among many others.
* Ionizing radiation such as the beta particles emitted by Lu-177 cause DNA damage to target cells through both direct and indirect mechanisms. In addition, ionizing radiation has also been shown to induce cell death through what is known as the bystander effect, a phenomenon where cellular signaling from irradiated cells towards non-irradiated cells induces cellular damage and eventually death in nearby surrounding cells.
* Lu-177-DOTATATE is a somatostatin analog that predominantly recognizes SSTR2. This reagent has been used extensively and its well-tolerated safety profile and efficacy has been shown in a variety of neuroendocrine tumors.

Primary Objective:

To assess the safety and to evaluate the ability of Lu-177-DOTATATE to improve upon progression-free survival (PFS) at 6 months in participants with inoperable, SSTR positive PHEO/PGL by comparing PFS of participants treated with Lu-177-DOTATATE to historical controls from existing literature.

Eligibility:

* Histologically-proven, surgically inoperable, PHEO/PGL participants (both newly diagnosed or participants with existing diagnoses are eligible)
* Must have presence of SSTR+ disease as documented by positive Ga-68-DOTATATE PET scan

  * Positivity of Ga-68-DOTATATE PET scan defined as having at least one lesion that is greater than or equal to 10 mm in diameter with uptake that is higher than or equal to liver and is qualitatively higher and distinguishable from background activity.
  * Measurable disease as defined by RECIST 1.1
* Age: greater than or equal to 18
* Karnofsky Performance Score greater than or equal to 60 or, ECOG Performance Status of 2 or better
* Able to understand and willing to sign informed consent

Design:

* Open-label, single-arm, multi-center, phase 2 study evaluating efficacy and safety of Lu- 177-DOTATATE in the selected participant population divided into two cohorts: 1) SDHx cohort will include participants with the succinate dehydrogenase mutation, which is the most common and most aggressive genetic sub-group of participants with PHEO/PGL, and 2) apparent sporadic cohort which will include participants without a clear genetic mutation.
* Lu-177-DOTATATE is administered IV every 8 (+/- 2) weeks, for a total of 4 administrations. Gamma whole-body planar and/or SPECT/CT imaging of Lu-177-DOTATATE will be obtained at 4 to 72-hours post-injection to confirm localization of treatment to intended targets (optional for participating sites). A CT/MRI for RECIST, Ga-68-DOTATATE and F-18-FDG PETs will be obtained post-2 administrations and post-4 administrations.
* All participants will be contacted by phone within a week after each Lu-177-DOTATATE and in-person every 4 weeks. After the end of treatment visit at week 32, participant will continue to be followed every 12 weeks until 3 years after the first Lu-177-DOTATATE administration. Follow-up visits may be conducted remotely or via telemedicine. After the 3 years, all participants will be contacted yearly until death to assess survival and disease status.
* Participants who have met the primary endpoint of having achieved a PFS of at least 6 months after the initial treatment course, may be eligible to receive further cycles of Lu-177-DOTATATE at the time of progression.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Surgically inoperable participants with clinical diagnosis of PHEO/PGL who also have demonstrated disease histologically consistent with pheochromocytoma or paraganglioma (preferably confirmed by research site pathology review if initial pathology was done outside of research site, but not mandatory)
* Progressive disease by RECIST 1.1 with or without symptoms within the last 12 months. NOTE: Untreated participants with existing histologic diagnoses are eligible if progression can be demonstrated
* PHEO/PGL that is not associated with any known susceptibility genetic mutations for PHEO/PGL except SDHx mutation (a.k.a. "apparent sporadic"), based on documented genetic testing results obtained prior to study enrollment. PHEO/PGL that is associated with non-SDHx mutations such as VHL, NF1, and RET will not be eligible for this study.
* Both metastatic and inoperable primary-only participants are eligible.
* Must have presence of SSTR+ disease as documented by positive Ga-68-DOTATATE PET scan within 12 weeks of anticipated treatment.

NOTE:

* Positivity of Ga-68-DOTATATE PET scan defined as having at least one lesion that is greater than or equal to 10 mm in diameter with uptake that is higher than or equal to liver and is qualitatively higher and distinguishable from background activity.
* Measurable disease as defined by RECIST 1.1

  * Age greater than or equal to 18
  * Karnofsky Performance Score greater than or equal to 60 or ECOG Performance Status of 2 or better.
  * Able to understand and willings to sign informed consent.
  * Ability and willingness to obtain all required scans per study schedule.
  * Negative serum pregnancy test for women of child-bearing potential. NOTE: A female is not of childbearing potential if a prior history of hysterectomy with bilateral oophorectomy or other procedure has rendered the participant surgically sterile, or >2 years since last menstruation.
  * Female participants of childbearing potential and male participants who are not surgically sterile or with female partners of childbearing potential must agree to use effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal gel) prior to study entry, for the duration of study participation, and for 4 months for male participants or 7 months for female participants (10 half-lives of Lu-177) after the last dose of Lu-177-DOTATATE.
  * Must have outside endocrinologist/medical oncologist who can follow the participant after receiving PRRT (NIH only requirement).
  * Patients with secreting tumors must be receiving adequate pharmacologic catecholamine blockade as determined by the treating physician.
  * Ineligible, unable to or unwilling to receive standard first line therapy for PHEO/PGL.

EXCLUSION CRITERIA:

* Creatinine clearance <50 mL/min calculated by the MDRD method, eventually confirmed by measured creatinine clearance (or measured glomerular filtration rate (GFR) using plasma clearance methods.
* Serum albumin less than or equal to 3.0 g/dL unless prothrombin time is within the normal range.
* Liver dysfunction as evidenced by Child s Class C Liver Disease or worse Alternatively, AST or ALT > 2.5 times institutional upper limit of normal (ULN) unless liver metastases are present, in which case up to 5 times ULN would be allowed.
* Hb < 8.0 g/dL; WBC < 2.0 x 10^9/L (or Absolute Neutrophil Count < 1000); Platelets < 100 x 10^9/L
* In participants with symptoms of congestive heart failure, New York Heart Association (NYHA) classification of grade III or IV
* Pregnancy or lactation.
* Prior anti-tumoral radionuclide therapy with unsealed sources. Prior therapy with sealed radioactive sources such as brachytherapy will be allowed.
* Prior local radiation therapy would be allowed as long as there is at least one non-irradiated index lesion.
* Known brain metastases, unless these metastases have been treated and stabilized for at least 24 weeks, prior to enrollment in the study. Patients with a history of brain metastases must have a head CT or MRI scan with contrast to document stable disease for at least 24 weeks prior to enrolment in the study.
* Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and proven no evidence of recurrence for 5 years.
* Patients who participated in any therapeutic clinical study with an investigational agent within the last 30 days.
* Patients may be on somatostatin analogue therapy (e.g. but not only limited to sandostatin or lanreotide therapy). However, therapy with somatostatin analogues should not be initiated or altered within 3 months of study enrolment. Patients on short term octreotide may have dose held for 24 hours prior to Lu-177-DOTATATE therapy. Those on long acting octreotide therapy will receive treatment at 1 to 5 days prior to their next cold octreotide dose, in order to prevent competition for the receptor.
* Patient weight > 400 lbs (table limit for PET scanner) or per local institutional standard for participating sites.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, hypertension (>180/110), arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Inability to tolerate at least one modality of diagnostic anatomic imaging, such as CT or MRI.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 6 months
  Median amount of time subject survives without disease progression after treatment

SECONDARY OUTCOMES:
Time to tumor progression | at disease progression
  Median amount of time subject survives without disease progression after treatment
Safety and tolerability profile | 30 days after the last dose of study drug
  List of adverse event frequency
Overall survival | at death
  Median amount of time subject survives after therapy
Objective response rate | at disease progression
  Proportion of patients whose tumors shrunk after therapy
Evaluate Quality of Life | 3 years
  Proportion of patients with increased Quality of Life (QoL)
Determine changes in plasma biochemical markers | 3 years
  changes in plasma biochemical markers
Determine ability to decrease anti-hypertensive medication | 3 years
  Proportion of patients using decreased amount of anti-hypertensive medication

CONTACTS AND LOCATIONS:
Overall Officials: Frank I Lin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Kim SJ, Pak K, Koo PJ, Kwak JJ, Chang S. The efficacy of (177)Lu-labelled peptide receptor radionuclide therapy in patients with neuroendocrine tumours: a meta-analysis. Eur J Nucl Med Mol Imaging. 2015 Dec;42(13):1964-70. doi: 10.1007/s00259-015-3155-x. Epub 2015 Aug 9. PMID 26253273
- [Background] Lenders JW, Duh QY, Eisenhofer G, Gimenez-Roqueplo AP, Grebe SK, Murad MH, Naruse M, Pacak K, Young WF Jr; Endocrine Society. Pheochromocytoma and paraganglioma: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2014 Jun;99(6):1915-42. doi: 10.1210/jc.2014-1498. PMID 24893135
- [Background] Maurice JB, Troke R, Win Z, Ramachandran R, Al-Nahhas A, Naji M, Dhillo W, Meeran K, Goldstone AP, Martin NM, Todd JF, Palazzo F, Tan T. A comparison of the performance of (6)(8)Ga-DOTATATE PET/CT and (1)(2)(3)I-MIBG SPECT in the diagnosis and follow-up of phaeochromocytoma and paraganglioma. Eur J Nucl Med Mol Imaging. 2012 Aug;39(8):1266-70. doi: 10.1007/s00259-012-2119-7. Epub 2012 Apr 20. PMID 22526961
- [Derived] Haque F, Carrasquillo JA, Turkbey EB, Mena E, Lindenberg L, Eclarinal PC, Nilubol N, Choyke PL, Floudas CS, Lin FI, Turkbey B, Harmon SA. An automated pheochromocytoma and paraganglioma lesion segmentation AI-model at whole-body 68Ga- DOTATATE PET/CT. EJNMMI Res. 2024 Nov 5;14(1):103. doi: 10.1186/s13550-024-01168-5. PMID 39500789
- [Derived] Gubbi S, Al-Jundi M, Auh S, Jha A, Zou J, Shamis I, Meuter L, Knue M, Turkbey B, Lindenberg L, Mena E, Carrasquillo JA, Teng Y, Pacak K, Klubo-Gwiezdzinska J, Del Rivero J, Lin FI. Early short-term effects on catecholamine levels and pituitary function in patients with pheochromocytoma or paraganglioma treated with [177Lu]Lu-DOTA-TATE therapy. Front Endocrinol (Lausanne). 2023 Oct 11;14:1275813. doi: 10.3389/fendo.2023.1275813. eCollection 2023. PMID 37886645
- [Derived] Gubbi S, Al-Jundi M, Del Rivero J, Jha A, Knue M, Zou J, Turkbey B, Carrasquillo JA, Lin E, Pacak K, Klubo-Gwiezdzinska J, Lin FI. Case Report: Primary Hypothyroidism Associated With Lutetium 177-DOTATATE Therapy for Metastatic Paraganglioma. Front Endocrinol (Lausanne). 2021 Jan 21;11:587065. doi: 10.3389/fendo.2020.587065. eCollection 2020. PMID 33551992
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-C-0087.html